CLINICAL TRIAL: NCT06618079
Title: A Two Cohort, Single-sequence, Parallel, Open Label, Multiple Oral Dosing Phase 1 Clinical Trial to Evaluate the Safety and the Pharmacokinetic Drug-drug Interaction of HUC2-565-A and HUC2-565-B in Healthy Adult Volunteers
Brief Title: Drug-Drug Interaction Study Between HUC2-565-A and HUC2-565-B
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUC2-565_P1_DDI
Record Dates: First submitted 2024-04-22; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Evaluate the effect of S-Amlodipine on the pharmacokinetic properties of Azilsartan under steady states.
  Interventions: Drug: HUC2-565-A, HUC2-565-A and HUC2-565-B
- Cohort B (Experimental): Evaluate the effect of Azilsartan on the pharmacokinetic properties of S-amlodipine under steady states.
  Interventions: Drug: HUC2-565-B, HUC2-565-A and HUC2-565-B

INTERVENTIONS:
Drug: HUC2-565-A, HUC2-565-A and HUC2-565-B — Cohort A received HUC2-565-A for 5 days, followed by HUC2-565-A and HUC2-565-B for 9 days.
  Arms: Cohort A
Drug: HUC2-565-B, HUC2-565-A and HUC2-565-B — Cohort B takes HUC2-565-B for 9 days, then HUC2-565-A and HUC2-565-B for 5 days.
  Arms: Cohort B

SUMMARY:
The purpose of this study is to evaluate a pharmacokinetic drug interaction and safety.

DETAILED DESCRIPTION:
Cohort A: To evaluate the effect of S-Amlodipine on the pharmacokinetics of Azilsartan at steady state.

Cohort B: To evaluate the effect of Azilsartan on the pharmacokinetics of S-Amlodipine at steady state.

ELIGIBILITY:
[ Inclusion Criteria ]

1. Healthy adult volunteer aged 19 years or older at the pre-study(screening)
2. Volunteer with a body mass index(BMI) of 18.0 kg/m2 or more and 30.0 kg/m2 or less, with a 50kg or more weight at the pre-study(screening)
3. A person who has no chronic disease requiring birth or treatment and has no pathological symptoms or findings as a result of medical examination
4. Volunteer who is judged to be suitable as a clinical trial subject as a result of screening test within 28 days of the first administration of the investigational product.
5. A person who, after hearing and fully understanding the details of this clinical trial, voluntarily decides to participate and agrees to comply with the compliance of the test subjects during the clinical trial period

[ Exclusion Criteria ]

1. Current or past medical history of the liver, kidney, nervous system, respiratory system, endocrine system, blood disease, tumor, Urogenital system, cardiovascular system, digestive system, musculoskeletal system, etc., which are clinically significant, in addition to current symptoms or past medical history.
2. Person with a history of gastrointestinal diseases(Crohn's disease, ulcers, acute or chronic pancreatitis) or gastrointestinal surgery(except for simple appendectomy or hernia surgery) that may affect Investigational product absorption
3. Pregnant women(Urine-HCG positive person) or breastfeeding mother
4. Person with a history of hypersensitivity(anaphylaxis or angioedema, etc) or clinically significant hypersensitivity reactions to drugs, formulation additives, and other drugs(aspirin, penicillin antibiotics, macrolide antibiotics, etc), including components Azilsartan and S-amlodipine
5. Those who have clinically significant findings, including the following findings on 12-lead electrocardiogram test(screening)

   * in case of men QTc > 450ms, in case of women QTc > 470ms
   * PR interval > 200ms
   * QRS duration > 120ms
6. Those who show clinically significant results on the clinical laboratory examination, including the following results(screening)

   * Those whose AST, ALT, ALP, r-GT and Bilirubin total exceed twice the upper limit of the normal range in the clinical laboratory test for liver function evaluation.
   * If the level of creatine in the blood is outside the reference range or the eGFR calculated by the CKD-EPI formula is less than 60mL/min/1.73m2
   * Those whose blood total cholesterol and LDL-cholesterol levels exceed 1.5 times the upper limit of the normal range
   * Clinical laboratory examination in which CPK exceeds 2.5 times the upper limit of the normal range
7. A person with a history of substance abuse or who has tested positive for substance abuse in a urine drug test.
8. A person whose blood pressure and pulse rate fall within the following range in the vital signs measured from the upper left after resting for at least 3 minutes during screening

   * systolic blood pressure ≥ 150 mmHg or ≤ 90mmHg
   * diastolic blood pressure ≥ 100 mmHg or ≤ 60mmHg
   * pulse ≤ 40 bpm ≥ 100 bpm
9. Food eaters who eat abnormal diets that may affect absorption, distribution, metabolism and excretion of investigational products or may affect drug metabolism
10. A person who has administered a prescription drug or herbal medicine that may affect the characteristics of the clinical trial drug within two weeks of the first administration of the clinical trial drug, or has administered a over the counter drug(OTC drug) or health functional food within two weeks. (However, if the drug does not affect the pharmacokinetic properties of the investigational products, it may participate in the clinical trial at the discretion of the investigator.)
11. A person who has taken drug metabolism enzyme induction and inhibitory drugs such as barbiturates drugs within one month prior to the first administration date of the investigational products.
12. A person who participated in other clinical trials and received the administration within 6 months prior to the first administration of the investigational products for clinical trials
13. A person who has donated whole blood within two months prior to the first administration of the investigational products, or has donated ingredients within one month, received a blood transfusion within one month, or is prohibited from donating blood from the time of written consent until the time of PSV
14. A person who has been drinking continuously(over 21 units/week, 1unit=10g=12.5mL of pure alcohol) within 6 months prior to the first administration date of the investigational products or who is unable to abstain from drinking from the time of written consent until the time of PSV
15. Smokers whose average daily amount of smoking exceeds 10 cigarettes within three months prior to the first administration date of clinical trials and those who are unable to quit smoking from 24 hours before the first administration to the last time of blood collection.
16. A person who has consumed or cannot prohibit the consumption of grapefruit-containing food from 48 hours before the first administration of the clinical trial drug to the time of PSV
17. A person who has consumed or cannot prohibit the consumption of caffeine-containing food(coffee, green tea, black tea, soda, coffee milk, nutritional tonic drink, etc) during the period from 24 hours before the first administration of the investigational products to the time of last blood collection
18. A person who has exercised intense exercise exceeding the standard of daily life or is forced to exercise intensely during the period from 48 hours before the first administration of clinical trials drugs to the time of PSV
19. A person who is not using a recognized contraceptive method(For example: Contraceptive administration and transplantation or intrauterine devices, fertility procedures (such as tubectomy, sphincter ligation), blocking methods (used in combination with condoms, contraceptive vaginal membranes, vaginal sponges or cervical caps)) even if he/she, his/her spouse, or his/her partner is planning to become pregnant or not until two weeks after the date of last clinical trial drug administration from the time of written consent
20. A person who is not suitable for participation in clinical trials due to other reasons other than the above inclusion/exclusion criteria at the discretion of the examiner

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
AUCtau,ss | 0-14days
  Pharmacokinetic parameter
Cmax,ss | 0-14days
  Pharmacokinetic parameter

SECONDARY OUTCOMES:
AUCinf,ss | 0-14days
  Pharmacokinetic parameter
Tmax,ss | 0-14days
  Pharmacokinetic parameter
T1/2,ss | 0-14days
  Pharmacokinetic parameter
CLss/F | 0-14days
  Pharmacokinetic parameter
Vdss/F | 0-14days
  Pharmacokinetic parameter
Cmin,ss | 0-14days
  Pharmacokinetic parameter
Cav,ss | 0-14days
  Pharmacokinetic parameter
PTF(Peak-to-trough fluctuation) | 0-14days
  Pharmacokinetic parameter
Metabolic ratio | 0-14days
  Pharmacokinetic parameter

CONTACTS AND LOCATIONS:
Overall Officials: Min Gyu Park, Principal Investigator — Chungbuk National University Hospital
Locations (1):
- Chungbuk national university hospital, Jungbuk, South Korea

IPD SHARING:
Plan to Share IPD: No